CLINICAL TRIAL: NCT05153928
Title: Management of Uterine Leiomyomata and Adenomyosis : Role of Hysteroscopy in Diagnosis and Norethisterone in the Treatment
Brief Title: Management of Uterine Leiomyomata and Adenomyosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ahmed Ali Mahmoud (Other)
Collaborators: Assiut University (Other)
Responsible Party: Sponsor-Investigator, Ahmed Ali Mahmoud, Dr, Assiut University
Organization: Assiut University (Other)
Other Study IDs: 12091984
Record Dates: First submitted 2021-11-30; First posted 2021-12-10 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-11

CONDITIONS: Abnormal Uterine Bleeding
MeSH Terms: conditions — Metrorrhagia | interventions — Norethindrone Acetate

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Histopathological study
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- fibroid cases: Norethisterone acetate for 5 months
  Interventions: Drug: Norethisterone acetate
- adenomyosis: Norethisterone acetate for 5 months
  Interventions: Drug: Norethisterone acetate

INTERVENTIONS:
Drug: Norethisterone acetate — Norethisterone acetate for 5 months

SUMMARY:
1. to determine the role of hysteroscopy and guided biopsy to differentiate between submucosal fibroids and adenomyosis confirmed by histopathological examination
2. to evaluate the efficacy of norethisterone in the treatment of symptomatic adenomyosis and leiomyoma

DETAILED DESCRIPTION:
The aim of the present study is:

1. to determine the role of hysteroscopy and guided biopsy to differentiate between submucosal fibroids and adenomyosis confirmed by histopathological examination
2. to evaluate the efficacy of norethisterone in the treatment of symptomatic adenomyosis and leiomyoma

ELIGIBILITY:
Inclusion Criteria:

- (1) age≥30 years; (4) dysmenorrhea, adenomyosis-associated chronic pain, and/or menorrhagia.

(3) regular menstrual cycles before administration of norethisterone; (4) no other treatment for adenomyosis/leiomyomatosis at least for 3 months biopsies and histopathology for operated patients;

Exclusion Criteria:

* (1) pregnant and/or breast-feeding women (2) patients with a ovarian neoplasm, benign ovarian cyst including endometrioma, pelvic inflammatory disease or other endocrine diseases.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: single arm single center study
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-04-10 (Actual); Primary Completion 2021-11-25 (Actual); Study Completion 2021-12-25 (Estimated)

PRIMARY OUTCOMES:
is to evaluate sensitivity and specificity of hysteroscopy in differentiating between uterine adenomyosis and leiomyomatosis | 6 months
  Symptomatic improvement

CONTACTS AND LOCATIONS:
Overall Officials: Hisham Mo Taleb, Md, Principal Investigator — Assiut University
Locations (2):
- Egypt (2):
  - Ahmed Ali, Asyut
  - Maternaty hospital in assiut, Asyut

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wilde S, Scott-Barrett S. Radiological appearances of uterine fibroids. Indian J Radiol Imaging. 2009 Jul-Sep;19(3):222-31. doi: 10.4103/0971-3026.54887. PMID 19881092